CLINICAL TRIAL: NCT03266120
Title: Assessing Human Health Benefits of Gardening
Brief Title: Health Benefits of Gardening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201701647
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Anxiety; Depression; Healthy; Mood Disturbance; Stress; Quality of Life; Physical Activity; Social Interaction
Keywords: Gardening; Therapeutic Arts; Therapeutic Horticulture; Anxiety; Depression; Mood States; Quality of Life; Social Interactions; Stress; Wellness
MeSH Terms: conditions — Anxiety Disorders; Depression; Motor Activity | interventions — Reproductive Techniques, Assisted; Gardening; Horticulture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Intervention (Active Comparator): Participants randomly assigned to this arm will receive a hands-on art intervention that will consist of twice weekly group sessions of approximately 60 minutes each in duration that will take place indoors over a period of four weeks for a total of eight art sessions. Participants will complete sets of self-report psychometric assessments and blood pressure and heart rate will be monitored before, during, and following the conclusion of the intervention.
  Interventions: Other: Art
- Gardening Intervention (Experimental): Participants randomly assigned to this arm will receive a hands-on gardening intervention that will consist of twice weekly group sessions of approximately 60 minutes each in duration that will take place in a greenhouse over a period of four weeks for a total of eight gardening sessions. Participants will complete sets of self-report psychometric assessments and blood pressure and heart rate will be monitored before, during, and following the conclusion of the intervention.
  Interventions: Other: Gardening

INTERVENTIONS:
Other: Art — Participants will receive a hands-on art activities intervention consisting of two art activities sessions each week lasting approximately 60 minutes each in duration for four weeks for a total of eight sessions. Art activities will include hand papermaking, image transfer, visual storytelling, linocut printmaking, paper batik, mixed media collage, and sensation drawing based activities. Participants will complete sets of self-report psychometric assessments before, during, and following the art intervention. Heart rate and blood pressure will be monitored before, during, and following completion of the art intervention.
  Arms: Art Intervention
Other: Gardening — Participants will receive a hands-on gardening intervention consisting of two gardening sessions each week lasting approximately 60 minutes each in duration for four weeks, for a total of eight sessions. Gardening activities will include planting seeds, bulbs and tubers, transplanting seedlings, vegetative propagation and sight, smell, taste and touch sensory based activities. Participants will complete sets of self-report psychometric assessments before, during, and following the gardening intervention. Heart rate and blood pressure will be monitored before, during, and following completion of the gardening intervention.
  Other Names: Horticulture; People-Plant Interactions
  Arms: Gardening Intervention

SUMMARY:
The objective of the research is to test the hypothesis that participating in group-based gardening or group-based art activities may alter the mental health and cardiac physiological status of a wellness population of women ages 26-49. Assessment of the effects of gardening or art activities on the experimental population will take two approaches, the first being the use of physiological measurements of heart rate and blood pressure. The second approach will employ six widely used and well-established self-reported assessment instruments that will capture information about the health and well-being of participants. These measurements and assessments will provide a psychometrically-based before and after mental health status and between treatments health summaries of the participants in the gardening group and those engaged in the art group activities.

DETAILED DESCRIPTION:
The goal of this project is to better understand how interacting and working with plants in a group gardening activities program in a greenhouse, or a group art program that takes place indoors and is devoid of images or depictions of plants influences the overall health and well-being of participants.

A total anticipated study population (N = 40) will consist of up to 20 healthy women randomly assigned to the art activities group, and up to 20 healthy women assigned to the gardening group. There will be measurements of heart rate, systolic and diastolic blood pressure, and psychometric assessments including satisfaction of social activities at baseline and post intervention. Heart rate and blood pressure measurements will be taken at the beginning and end of each of the eight gardening or arts sessions. Psychometric assessments of study participants will be conducted at baseline and post-intervention. Each treatment group will be divided into two smaller groups of up to ten women each that will receive the gardening or art interventions on different days of the week. The participants in the gardening or art groups will receive an experimental intervention consisting of 8 gardening or art sessions, each approximately 60 minutes in duration over a four week treatment period. Gardening and art sessions will take place at the same time of day twice each week, and follow a standardized programming sequence to ensure equivalency of intervention across all sessions. Ambient environmental conditions in the greenhouse during the gardening sessions will be monitored and recorded. The gardening activities will emphasize growing plants from seeds, plant propagation techniques, transplanting, and plant-mediated taste, visual, olfactory and touch sensory stimulation. All gardening sessions will begin with a short educational module introducing the plants and gardening activities taking place during each session. Art activities will include papermaking, image transfer, visual storytelling, linocut printmaking, paper batik, mixed media collage, and sensation drawing, and begin with a short educational module of the activity.

In addition to the pre- and post-intervention assessments and measurement, psychometric assessments will be administered for depression symptomatology, mood states and perceived stress at specific points during the gardening and art activities to evaluate any changes over time resulting from the interventions. Participant heart rate and blood pressure measurements will be made at the beginning and at the end of all gardening and art sessions.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* 26 - 49 years of age
* Not pregnant
* Non-gardener
* Non-artist
* Non-smoker
* Good Health
* Able to participate in all aspects of the study, including working with plants.

Exclusion Criteria:

* Uncomfortable in close spaces (claustrophobia)
* Allergies to plants
* Allergies to plant parts like pollen
* Allergies to plant-based foods
* No additions to alcohol or to recreational drugs or prescription medications
* Not suffering from recurring pain, and
* No diseases, disorders or disabilities that affect daily life.

Ages: 26 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2017-11-09 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Biometric Changes in Heart Rate | Baseline, up to 5 weeks
  Heart rate will be monitored using a portable electronic wrist cuff monitor. Participant heart rate will be measured at the beginning and end of each Individual treatment session, and before the beginning and after the completion of the entire treatment interventions.
Biometric Changes in Blood Pressure | Baseline, up to 5 weeks
  Blood pressure will be monitored using a portable electronic wrist cuff blood pressure monitor that records systolic and diastolic pressure. Participant blood pressure measurements will be recorded before and after each individual treatment session, and before the beginning and after the completion of the entire treatment interventions.

SECONDARY OUTCOMES:
Biometric Changes in Overall Health Status | Baseline, up to 5 weeks
  The SF-36v2 Health Survey assessment instrument (Ware and Sherbourne 1992; Hays et al 1993) will be used to evaluate eight scales that link to physical and mental health over a 4-week recall interval. This will reveal whether engaging in gardening activities will or will not result in changes in the overall health status based on instrument's physical and mental health subcomponent assessments of the gardening treatment group compared to the control group. The overall assessment scale for the SF-36 ranges from a low of 36 to a high of 400, with the U.S. norm being 314.
Biometric Changes in Depressive Symptomatology | Baseline, up to 5 weeks
  The study protocol will use the Beck Depression Inventory 2nd edition (BDI-II) (Beck et al 1988) with a recall interval of 2-weeks to gain insight relative to the intensity of depression. This assessment will determine whether engaging in gardening will or will not result in changes in depressive symptomatology of the gardening treatment group relative to the control group. The assessment scale for the Beck BDI ranges from a low of 10 to a high of 63. Scores 0-13 indicate minimal depressive symptomatology and above 19 up to 63 moderate to severe depressive symptomatology.
Biometric Changes in State Anxiety | Baseline, up to 5 weeks
  The State Trait Anxiety Inventory (STAI) instrument (Form Y) (Spielberger et al 1983) will be used in this study to gain insight regarding the relative intensity of anxiety being experienced by the gardening treatment group relative to the control group. The STAI reports on "at this moment" status. The STAI assessment will seek to determine whether engaging in gardening will or will not result in changes in State Anxiety status of the participants. The overall assessment scale for the STAI-Y ranges from a low of 20 to a high of 80, with higher scores indicating greater intensity of anxiety.
Biometric Changes in Mood States | Baseline, up to 5 weeks
  The study protocol will employ the Profile of Mood States 2nd edition short form for adults instrument (POMS2-AS) with an immediate recall interval (McNair et al 1981; Shacham 1983) to gain insight of the relative to transient and fluctuating moods and enduring states of affect. The POMS2-AS will assess whether engaging in gardening activities will or will not result in changes in mood and enduring states of affect status of the gardening treatment group relative to the control group, both during and following the completion of the gardening activities treatment regimen. The assessment scale for the POMS2-AS ranges from 5 to a high of 100 per scale .
Biometric Changes in Perceived Stress | Baseline, up to 5 weeks
  The study will use the Perceived Stress Scale (PSS) (Cohen et al 1983) with a recall interval of 4-weeks to gain insight relative to the intensity of perceived stress. This assessment will determine whether engaging in gardening activities will or will not result in changes in the perceived stress levels of the gardening treatment group relative to the control group. The assessment scale for the Perceived Stress Scale ranges from a low of 0 to a high of 40, indicating higher stress at higher scores. The norm score for women is 13.7.
Biometric Changes in Satisfaction in Social Activities | Baseline, up to 5 weeks
  The study will use the The Satisfaction with Participation in Discretionary Social Activities (SPDSA) PROMIS short form v1.0 instrument to assess contentment with participants' leisure time and affairs with friends, and encompasses a recall interval of one week (Hahn et al 2010)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Guy, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Fifield and Merhof Halls, Gainesville, Florida
  - Wilmot Gardens Conference Center and Greenhouse, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Beck, AT, Steer RA, Garbin MG. Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clinical Psychology Review 1988 (8):77-100.
- [Background] Spielberger, CD, Gorsuch RL, Lushene R. The State-Trait Personality Inventory STAI-Y, form Y. Consulting Psychologists Press, Palo Alto. 1983
- [Background] McNair PM, Lorr M, Droppleman LF. POMS manual (2nd ed.). San Diego: Educational and Industrial Testing Service. 1981.
- [Background] Shacham S. A shortened version of the Profile of Mood States. J Pers Assess. 1983 Jun;47(3):305-6. doi: 10.1207/s15327752jpa4703_14. PMID 6886962
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Hahn EA, Beaumont JL, Pilkonis PA, Garcia SF, Magasi S, DeWalt DA, Cella D. The PROMIS satisfaction with social participation measures demonstrated responsiveness in diverse clinical populations. J Clin Epidemiol. 2016 May;73:135-41. doi: 10.1016/j.jclinepi.2015.08.034. Epub 2016 Feb 27. PMID 26931288
- [Derived] Odeh R, Diehl ERM, Nixon SJ, Tisher CC, Klempner D, Sonke JK, Colquhoun TA, Li Q, Espinosa M, Perdomo D, Rosario K, Terzi H, Guy CL. A pilot randomized controlled trial of group-based indoor gardening and art activities demonstrates therapeutic benefits to healthy women. PLoS One. 2022 Jul 6;17(7):e0269248. doi: 10.1371/journal.pone.0269248. eCollection 2022. PMID 35793277